CLINICAL TRIAL: NCT01240304
Title: A Phase II Study to Assess the Efficacy and Safety of Preoperative Chemotherapy With Radiation Therapy for Patients With Borderline Unresectable Adenocarcinoma of the Pancreas
Brief Title: A Phase II Study to Assess the Efficacy and Safety of Preoperative Chemo With Radiation Therapy for Patients With Borderline Unresectable Adenocarcinoma of the Pancreas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no subjects enrolled
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112748
Record Dates: First submitted 2010-11-09; First posted 2010-11-15 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiotherapy; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine, radiation therapy, surgery (Experimental)
  Interventions: Drug: Gemcitabine; Radiation: Radiation therapy; Procedure: pancreaticoduodenectomy

INTERVENTIONS:
Drug: Gemcitabine — The course of preoperative treatment in this study will consist of an alternating combination of 6mg/M² of Gemcitabine for 24 hours and 7.0 Gy (radiation) of radiation therapy. The subject will undergo one of these therapies alternating daily for a total of 10 days then the subject will be allowed to rest for 4 weeks before undergoing restaging and surgery. After surgery, the subject will then undergo the conventional chemotherapy regimen consisting of 6 cycles (1 cycle = 28 days) of 1000mg/M² of Gemcitabine over a 30 minute infusion rate.
  Other Names: Gemzar
Radiation: Radiation therapy — The course of preoperative treatment in this study will consist of an alternating combination of 6mg/M² of Gemcitabine for 24 hours and 7.0 Gy (radiation) of radiation therapy. The subject will undergo one of these therapies alternating daily for a total of 10 days then the subject will be allowed to rest for 4 weeks before undergoing restaging and surgery. After surgery, the subject will then undergo the conventional chemotherapy regimen consisting of 6 cycles (1 cycle = 28 days) of 1000mg/M² of Gemcitabine over a 30 minute infusion rate.
Procedure: pancreaticoduodenectomy — Surgery will be planned 28 days (+/- 3 days) after the last dose of chemotherapy. The liver and pancreas will be examined by palpation and inspection. In the absence of metastases, tumor mobilization and surgical resection will be performed with standard surgical technique.
  Other Names: Removal of pancreas

SUMMARY:
The purpose of this phase II clinical trial study is to assess the resection rate among subjects who have been initially diagnosed with unresectable or borderline resectable pancreatic adenocarcinoma. This will be done by providing preoperative treatment that will include alternating cycles of chemotherapy and radiotherapy treatment. In addition, this clinical trial will assess the safety of preoperative chemotherapy with radiation therapy for subjects with unresectable or borderline resectable adenocarcinoma of the pancreatic head, assess margin-negative resection rates, disease-free survival, assess overall survival rates, and determine patterns of local and distant recurrence.

DETAILED DESCRIPTION:
The purpose of this phase II clinical trial study is to assess the resection rate among subjects who have been initially diagnosed with unresectable or borderline resectable pancreatic adenocarcinoma. This will be done by providing preoperative treatment that will include alternating cycles of chemotherapy and radiotherapy treatment. In addition, this clinical trial will assess the safety of preoperative chemotherapy with radiation therapy for subjects with unresectable or borderline resectable adenocarcinoma of the pancreatic head, assess margin-negative resection rates, disease-free survival, assess overall survival rates, and determine patterns of local and distant recurrence.

The study population in this clinical trial will consist of untreated subjects 18 years or older who have a histologically or cytologically confirmed diagnosis of unresectable or borderline resectable adenocarcinoma of the pancreatic head. Once the patient has undergone the necessary tests and the tumor has been staged, the principal investigator or co-investigators will determine if the patient is suitable to be inducted in this clinical trial. The course of preoperative treatment in this study will consist of an alternating combination of 6mg/M² of Gemzar for 24 hours and 7.0 Gy of radiation therapy. The subject will undergo one of these therapies alternating daily for a total of 10 days then the subject will be allowed to rest for 4 weeks before undergoing restaging and surgery. After surgery, the subject will then undergo the conventional chemotherapy regimen consisting of 6 cycles of 1000mg/M² of Gemzar over a 30 minute infusion rate.

The primary outcome of this clinical trial is the margin-negative resection rate. This will be determined by the tumor's response to the pre/post-operative treatment so that the tumor can be removed surgically via pancreaticoduodenectomy. Once the subject has completed the treatment as described in the protocol, he/she will continued to be followed to assess survival and patterns of local and distance recurrence. The purpose of this clinical trial will be an attempt to provide subjects with a more hopeful alternative to treatment for a disease that otherwise offers a grim prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 years and above. There will be no upper age restriction.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2. (See Appendix A -ECOG Performance Status Scale).
3. Cytologic or histologic proof of adenocarcinoma of pancreas.
4. Adequate renal, and bone marrow function:

   1. Leukocytes >= 3,000/uL (upper limit)
   2. Absolute neutrophil count >= 1,500/uL (upper limit)
   3. Platelets >= 100,000/Ul
   4. Serum creatinine <= 2.0 mg/dL
5. Hepatic function (endoscopic or percutaneous drainage as needed)

   a. Aspartate aminotransferase (AST)-(SGOT)/Alanine aminotransferase (ALT) (SGPT) <= 5 X institutional ULN (upper limit of normal)
6. Borderline resectable pancreatic cancer:

   1. Short segment hepatic artery abutment (< 180° involvement)
   2. Tumor abutment (<180° ) of superior mesenteric artery
   3. Superior mesenteric/portal vein involvement beyond that of a simple resection and reconstruction
   4. Pancreatitis that obscures the determination of vessel involvement and may preclude an otherwise curative operation
7. Unresectable pancreatic cancer:

   1. Tumors that encase (> 180° involvement) single or multiple arteries and veins (celiac axis, superior mesenteric artery, superior mesenteric/portal vein, hepatic artery)
   2. Occlusion of superior mesenteric/portal vein

Exclusion Criteria:

1. Infections such as cholangitis, pneumonia, or wound infections that would preclude protocol therapy.
2. Women with a positive urine or serum pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to refrain from breast feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence.
3. Subjects cannot have known heptic or peritoneal metastases detected by ultrasound (US), CT scan, or laparotomy/laparoscopy prior to treatment.
4. Subjects with unstable angina or New York Heart Association (NYHA) Grade II or greater congestive heart failure will be excluded (see Appendix B).
5. Known presence of central nervous system or brain metastases
6. Subjects with prior radiotherapy to the upper abdomen or liver will be excluded.
7. Subjects will be excluded if deemed unable to comply with study and/or follow-up procedures.
8. Subjects with a known hypersensitivity to Gemzar are excluded.
9. Multiple positive lymph nodes, which will make the radiotherapy treatment volume too large. Peripancreatic involved nodes can be included in the radiotherapy treatment volume if the field of involved nodes is less than 7.5cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam Makhoul, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine, Radiation Therapy, Surgery: Alternating combination of 6mg/M² of Gemcitabine for 24 hours and 7.0 Gy (radiation) of radiation therapy. The subject will undergo one of these therapies alternating daily for a total of 10 days then the subject will be allowed to rest for 4 weeks before undergoing restaging and surgery. After surgery, the subject will then undergo the conventional chemotherapy regimen consisting of 6 cycles (1 cycle = 28 days) of 1000mg/M² of Gemcitabine over a 30 minute infusion rate.
  Radiation therapy: The course of preoperative treatment in this study will consist of an alternating combination of 6mg/M² of Gemcitabine for 24 hours and 7.0 Gy (radiation) of radiation therapy. The subject will undergo one of these therapies alternating daily for a total of 10 days then the subject will be allowed to rest for 4 weeks before undergoing restaging and surgery. After surgery, the subject will then undergo the convention
Period: Overall Study
Arm/Group | Gemcitabine, Radiation Therapy, Surgery
Started | 10
Completed | 0
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Radiation Therapy, Surgery
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Margin-negative Resection Rate
Description: This will be determined by the tumor's response to the pre/post-operative treatment so that the tumor can be removed surgically.
Time Frame: An average of 6 years
Population: Early termination. No subject completed study. No data collected. No data analysis was completed.
Arm/Group | Gemcitabine, Radiation Therapy, Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Gemcitabine, Radiation Therapy, Surgery
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Radiation Therapy, Surgery (N=10)
abdominal pain (Gastrointestinal disorders) | 1 (1)
nausea/vomiting (Gastrointestinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT01240304/Prot_SAP_000.pdf